CLINICAL TRIAL: NCT00588666
Title: Phase II Trial of Gemcitabine, Carboplatin, and Bevacizumab in Chemotherapy Naive Patients With Advanced/Metastatic Urothelial Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-006
Record Dates: First submitted 2007-12-26; First posted 2008-01-08 (Estimated); Results first posted 2016-01-22 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2015-12

CONDITIONS: Myeloproliferative Disorder; Urothelial Carcinoma; Cancer
Keywords: Myeloproliferative Disorder; urinary bladder; Cancer; ureter; renal pelvis; chemotherapy
MeSH Terms: conditions — Myeloproliferative Disorders; Carcinoma, Transitional Cell; Neoplasms | interventions — Bevacizumab; Carboplatin; Gemcitabine

ARMS (1):
- Bevacizumab, Carboplatin, Gemcitabine (Experimental): Patients will initially receive bevacizumab 10 mg/kg followed by a 2 week treatment-free interval. Treatment will then begin with combination therapy. Gemcitabine 1000 mg/m2 will be administered intravenously on day 1 and 8 and carboplatin AUC 4.5 on day 1 with treatment recycled every 21 days. Bevacizumab will be administered at a dose of 15 mg/kg on day 1 of each 21-day cycle. Restaging evaluations will be performed after every 3 cycles of treatment (approximately 9 weeks). Patients will receive a total of 6 cycles of chemotherapy unless disease progression or unacceptable toxicity occurs. Patients who achieve stable disease, a partial response, or a complete response after completion of 6 cycles, will be eligible to continue bevacizumab at the same dose and schedule until disease progression for a maximum of 18 additional doses.
  Interventions: Drug: Bevacizumab; Drug: Carboplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Bevacizumab
Drug: Carboplatin
Drug: Gemcitabine

SUMMARY:
Gemcitabine and carboplatin are two standard chemotherapy drugs used to treat tumors of the urothelial tract. These drugs do not shrink tumors in all patients and when they do, it is generally for a limited amount of time. This has led scientists to look for different ways to treat cancer.

New drugs have been developed to treat cancer that work differently than standard chemotherapy drugs. One new class of drugs are called 'angiogenesis-inhibitors'. These drugs attempt to decrease the blood supply to tumors. By doing so, this may limit the tumor's source of oxygen and nutrients and prevent the tumor from growing. Bevacizumab is an anti-angiogenic drug.

In some other cancers such as colon cancer and lung cancer, combining bevacizumab with standard chemotherapy shrinks tumors in a greater proportion of patients and makes patients live longer than using standard chemotherapy alone. This has never been tested in urothelial cancer and we do not know if bevacizumab will have the same effects in this disease. The purpose of this study is to find out what effects, good and/or bad, the combination of gemcitabine, carboplatin, and bevacizumab has on you and your cancer.

DETAILED DESCRIPTION:
This is a phase II trial of gemcitabine, carboplatin, and bevacizumab in chemotherapy naïve patients with advanced/metastatic transitional cell carcinoma (TCC) of the urothelial tract.

ELIGIBILITY:
Inclusion Criteria:

* Histologic documentation: diagnosis of transitional cell carcinoma of the bladder,urethra, ureter, or renal pelvis.
* Unresectable or metastatic disease
* Ineligible for cisplatin (or incurable with cisplatin)
* ≥ 4 weeks since prior RT
* Karnofsky Performance Status ≥ 60%
* Age ≥ 18 years of age
* Required Initial Laboratory Values: Absolute neutrophil count ≥ 1.2 x 109/L; Platelets ≥ 100 x 109/L; Bilirubin ≤ 1.5 times the upper limit of normal (x ULN) for the institution; Aspartate transaminase (AST) and alanine transaminase(ALT) ≤ 3.0 x ULN;Serum creatinine < 2.0 or calculated creatinine clearance (CrCl) ≥ 30 mL/min

Exclusion Criteria:

* Prior treatment with systemic chemotherapy (prior intravesical therapy is permitted)
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than a Genentech-sponsored bevacizumab cancer study
* Blood pressure of >150/100 mmHg
* Unstable angina
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* History of myocardial infarction within 6 months
* History of stroke within 6 months
* Clinically significant peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Presence of central nervous system or brain metastases
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0
* Anticipation of need for major surgical procedure during the course of the study
* Minor surgical procedures such as fine needle aspirations or core biopsies within 7 days prior to Day 0
* Pregnant (positive pregnancy test) or lactating
* Albuminuria as demonstrated by a urinary albumin of greater or = to 1.0 g/24 hr at screening
* History of abdominal fistula, gastrointestinal perforation, or intra abdominal abscess within 6 months prior to Day 0
* Serious, non-healing wound, ulcer, or bone fracture
* Inability to comply with study and/or follow-up procedures
* History of persistent gross hematuria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2006-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dean Bajorin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memorial Sloan-Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memoral Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan-Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center at Mercy Medical Center, Rockville Centre, New York
  - Memoral Sloan Kettering Cancer Center@Phelps, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan-Kettering web site — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Bevacizumab, Carboplatin, Gemcitabine: Patients will initially receive bevacizumab 10 mg/kg followed by a 2 week treatment-free interval. Treatment will then begin with combination therapy. Gemcitabine 1000 mg/m2 will be administered intravenously on day 1 and 8 and carboplatin AUC 4.5 on day 1 with treatment recycled every 21 days. Bevacizumab will be administered at a dose of 15 mg/kg on day 1 of each 21-day cycle. Restaging evaluations will be performed after every 3 cycles of treatment (approximately 9 weeks). Patients will receive a total of 6 cycles of chemotherapy unless disease progression or unacceptable toxicity occurs. Patients who achieve stable disease, a partial response, or a complete response after completion of 6 cycles, will be eligible to continue bevacizumab at the same dose and schedule until disease progression for a maximum of 18 additional doses.
Period: Overall Study
Arm/Group | Treatment
Started | 51
Completed | 47
Not Completed | 4
Not completed — Adverse Event | 4

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 37
Region of Enrollment [Number; unit: participants]
  United States | 51

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Time to Disease Progression
Description: Response and progression will be evaluated in this study using the international criteria by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee [JNCI, 92(3):205-216, 2000]. Changes in only the largest diameter (uni-dimensional measurement) are used in the RECIST criteria.
Time Frame: 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment
Number analyzed (Participants) | 47
months
  Time to Progression | 6.5 [4.7 to 7.8]
  Overall Survival | 13.9 [11.9 to 18.1]

2. Secondary Outcome: The Response Rate of Combination Therapy With Bevacizumab, Gemcitabine, and Carboplatin in Patients With Advanced/Metastatic TCC.
Time Frame: 3 years
Measure: Number; unit: percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 47
percentage of participants | 49

ADVERSE EVENTS:
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 29/51
Other Adverse Events (participants affected / at risk) | 15/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=51)
Myocardial ischemia (Cardiac disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Death (General disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Hemorrhage/Bleeding, other (General disorders) | 1 (1)
Hepatobiliary disease (Hepatobiliary disorders) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bladder infection (Infections and infestations) | 2 (2)
Tooth infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
Lipase increased (Investigations) | 1 (1)
Injury, poisoning, and procedural complications-other, specify-device complication (Injury, poisoning and procedural complications) | 2 (2)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neutrophil count decrease (Investigations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Platelet count decrease (Investigations) | 2 (3)
Renal and urinary disorders-other, specify-Renal failure (Renal and urinary disorders) | 3 (3)
Syncope (Nervous system disorders) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 8 (8)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=51)
Fatigue (General disorders) | 11 (30)
Nausea (Gastrointestinal disorders) | 3 (6)
Thrombosis/thrombus/embolism (Vascular disorders) | 4 (4)
Weight loss (Investigations) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes